CLINICAL TRIAL: NCT02472145
Title: A Randomized Phase 2/3 Study of DACOGEN® (Decitabine) Plus Talacotuzumab (JNJ-56022473; Anti CD123) Versus DACOGEN (Decitabine) Alone in Patients With AML Who Are Not Candidates for Intensive Chemotherapy
Brief Title: An Efficacy and Safety Study of Decitabine (DACOGEN) Plus Talacotuzumab (JNJ-56022473; Anti CD123) Versus Decitabine (DACOGEN) Alone in Participants With Acute Myeloid Leukemia (AML) Ineligible for Intensive Chemotherapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR107273; 56022473AML2002 (Other: Janssen Research & Development, LLC); 2015-001611-12 (EudraCT Number)
Record Dates: First submitted 2015-04-29; First posted 2015-06-15 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Leukemia, myeloid, acute; DACOGEN; Decitabine; JNJ-56022473; CLS362
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Decitabine plus Talacotuzumab (Experimental): Part A: For Cycle 1 of Part A, participants will receive talacotuzumab on Day 1. Starting from Cycle 2 of Part A, participants may receive decitabine on Day 1, 2, 3, 4, and 5, and talacotuzumab on Day 8 and 22 of a 28-day cycle.
  Part B Arm 1: Participants will receive decitabine on Day 1, 2, 3, 4, and 5, and talacotuzumab on Day 8 and 22 of a 28-day cycle.
  Interventions: Drug: Decitabine 20 mg/m^2; Drug: Talacotuzumab 9 mg/kg
- Decitabine (Active Comparator): Participants in Part B Arm 2 will receive decitabine on Day 1,2, 3, 4 and 5 of a 28-day cycle.
  Interventions: Drug: Decitabine 20 mg/m^2

INTERVENTIONS:
Drug: Decitabine 20 mg/m^2 — Decitabine 20 milligram per square meter (mg/[m^2]) from Day 1, 2, 3, 4 and 5 of a 28-day cycle.
  Other Names: DACOGEN
Drug: Talacotuzumab 9 mg/kg — Talacotuzumab 9 milligram per kilogram mg/kg on Day 8 and 22 of a 28-day cycle.
  Other Names: CSL362
  Arms: Decitabine plus Talacotuzumab

SUMMARY:
The primary objective of study Part A is to assess the safety of talacotuzumab (formerly CSL362) monotherapy and confirm the recommended Phase 2 dose (RP2D) in participants with acute myeloid leukemia (AML) for whom experimental therapy is appropriate. The primary objective of study Part B are to assess complete response (CR) rate and overall survival (OS) in participants with AML who are not eligible for intense induction chemotherapy and who are randomly assigned to receive decitabine plus talacotuzumab at the RP2D or decitabine alone.

DETAILED DESCRIPTION:
This is a 2-part, open-label, multicenter, Phase 2/3 study conducted in participants with AML who are suitable for experimental therapy (Part A) and in participants with untreated AML who are not eligible for intense induction chemotherapy or hematopoeitic stem cell transplantation (HSCT) (Part B). In Study Part A, the safety, pharmacokinetic (PK) and pharmacodynamic (PD) profile will be assessed to confirm the RP2D of 9 milligram per kilogram (mg/kg) talacotuzumab. In Study Part B, participants will be randomized in a 1:1 ratio into either decitabine + talacotuzumab (arm 1) or decitabine alone (arm 2). Blood and bone marrow sampling will be done in Part A and B for disease assessment, PK, PD, and biomarkers will be collected in all participants. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* De novo or secondary acute myeloid leukemia (AML) (post myelodysplastic syndrome [MDS] or myeloproliferative neoplasm [MPN] or after leukemogenic chemotherapy) according to WHO 2008 criteria

For Part A:

- Participants With AML: treatment naive or relapsed for whom experimental therapy is appropriate (as assessed by their treating physician)

For Part B:

* Greater than or equal to (>=) 75 years of age or >= 65 up to 75 years of age and have at least one of the following: congestive heart failure or ejection fraction less than or equal to (<=) 50 percent; creatinine greater than (>) 2 milligram per deciliter (mg/dL); dialysis or prior renal transplant; documented pulmonary disease with lung diffusing capacity for carbon monoxide (DLCO) <= 65 percent of expected, or forced expiratory volume in 1 second (FEV1) <= 65 percent of expected or dyspnea at rest requiring oxygen; eastern cooperative oncology group (ECOG) performance status of 2; prior or current malignancy that does not require concurrent treatment; unresolved infection; comorbidity that, in the Investigator's opinion, makes the participant unsuitable for intensive chemotherapy and must be documented and approved by the Sponsor before randomization
* Previously untreated AML (except: emergency leukopheresis and/or hydroxyurea during the screening phase to control hyperleukocytosis but must be discontinued at least one day prior to start of study therapy)
* Not eligible for an allogeneic hematopoietic stem cell transplantation
* ECOG Performance Status score of 0, 1 or 2
* A woman must be either: Not of childbearing potential: postmenopausal (more than [>] 45 years of age with amenorrhea for at least 12 months; If, of childbearing potential must be practicing a highly effective method of birth control
* A woman of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) or urine pregnancy test at screening
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control eg, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository for at least 3 months after last study treatment

Exclusion Criteria:

* Acute promyelocytic leukemia with t(15;17), or its molecular equivalent (PML-RARalpha)
* For Part B only: Known leukemic involvement or clinical symptoms of leukemic involvement of the central nervous system
* Participants who received prior treatment with a hypomethylating agent
* For Part A only: Participants who did not recover from all clinically significant toxicities (excluding alopecia and hematologic toxicities) of any previous surgery, radiotherapy, targeted therapy, or chemotherapy to less than or equal to Grade 1
* Any uncontrolled active systemic infection that requires treatment with intravenous (IV) antibiotics
* A history of human immunodeficiency virus (HIV) antibody positive or tests positive for HIV if tested at screening
* Active systemic hepatitis infection requiring treatment or other clinically active liver disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 326 (Actual)
Dates: Start 2015-08-04 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (81):
- United States (11):
  - Orange, California
  - Aurora, Colorado
  - New Orleans, Louisiana
  - Detroit, Michigan
  - Lebanon, New Hampshire
  - New York, New York
  - Rochester, New York
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
- Australia (5):
  - Herston
  - Melbourne
  - Perth
  - South Woodville
  - Woolloongabba
- Belgium (7):
  - Antwerp
  - Hasselt
  - Leuven
  - Liège
  - Mons
  - Turnhout
  - Wilrijk
- France (7):
  - Grenoble
  - Lyon
  - Marseille
  - Montpellier
  - Nantes
  - Paris
  - Toulouse
- Germany (9):
  - Dresden
  - Düsseldorf
  - Essen
  - Frankfurt am Main
  - Hamburg
  - München
  - Münster
  - Ulm
  - Würzburg
- Israel (4):
  - Haifa
  - Jerusalem
  - Ramat Gan
  - Tel Aviv
- Poland (5):
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Warsaw
- Russia (7):
  - Chelyabinsk
  - Dzerzhinsk
  - Moscow
  - Nizhny Novgorod
  - Ryazan
  - Samara
  - Yekaterinburg
- South Korea (4):
  - Busan
  - Daegu
  - Hwasun Gun
  - Seoul
- Spain (7):
  - Badalona, Barcelona
  - Barcelona
  - Madrid
  - Pozuelo de Alarcon, Madrid
  - Salamanca
  - Seville
  - Valencia
- Sweden (4):
  - Gothenburg
  - Örebro
  - Stockholm
  - Uppsala
- Taiwan (4):
  - Chiayi City
  - Taichung
  - Tainan
  - Taipei
- Turkey (Türkiye) (4):
  - Ankara
  - Atakum
  - Istanbul
  - Izmir
- United Kingdom (3):
  - Bournemouth
  - Cardiff
  - Wolverhampton

REFERENCES:
- [Derived] Peipert JD, Efficace F, Pierson R, Loefgren C, Cella D, He J. Patient-reported outcomes predict overall survival in older patients with acute myeloid leukemia. J Geriatr Oncol. 2022 Sep;13(7):935-939. doi: 10.1016/j.jgo.2021.09.007. Epub 2021 Sep 11. PMID 34521609

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Decitabine + JNJ-56022473: Participants received 1 dose of JNJ-56022473 (talacotuzumab) at 9 milligram per kilogram (mg/kg) as intravenous (IV) infusion on Day 1 of cycle 1. From cycle 2 onwards, participants received decitabine 20 milligram per meter square (mg/m^2) IV on Day 1 to Day 5 followed by 9 mg/kg JNJ-56022473 on Day 8 and Day 22 of a 28-day cycle until treatment failure, relapse from complete response/remission (CR) or complete response with incomplete recovery (CRi), unacceptable toxicity, or death.
- Part B: Decitabine (Alone): Participants received decitabine 20 mg/m^2 IV on Days 1 to 5 of each 28-day cycle until treatment failure, relapse from CR or CRi, unacceptable toxicity, or death.
- Part B: Decitabine + JNJ-56022473: Participants received decitabine 20 milligram per meter square (mg/m^2) IV on Day 1 to Day 5 followed by 9 mg/kg JNJ-56022473 on Day 8 and Day 22 of a 28-day cycle until treatment failure, relapse from complete response/remission (CR) or complete response with incomplete recovery (CRi), unacceptable toxicity, or death.
Period: Overall Study
Arm/Group | Part A: Decitabine + JNJ-56022473 | Part B: Decitabine (Alone) | Part B: Decitabine + JNJ-56022473
Started | 10 | 159 | 157
Treated | 10 | 156 | 156
Safety | 10 | 165 (9 participants who received decitabine,not JNJ-56022473 included,3 untreated participant excluded.) | 147 (1 participant who was not treated and 9 participants who received only decitabine were excluded.)
Completed | 0 | 0 | 0
Not Completed | 10 | 159 | 157
Not completed — Death | 10 | 101 | 99
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 9 | 13
Not completed — Sponsor decision | 0 | 3 | 2
Not completed — Other | 0 | 45 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Decitabine + JNJ-56022473 | Part B: Decitabine (Alone) | Part B: Decitabine + JNJ-56022473 | Total
Number analyzed (Participants) | 10 | 159 | 157 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (10.88) | 75 (5.6) | 75.2 (5.32) | 74.8 (5.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 68 | 77 | 149
  Male | 6 | 91 | 80 | 177
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 5 | 9
  Not Hispanic or Latino | 10 | 143 | 143 | 296
  Unknown or Not Reported | 0 | 12 | 9 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All participants randomized into the study, grouped per treatment assigned by randomization, regardless of the actual treatment received. Here, 'N' (number of participant analyzed) signifies number of participants who were evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 10 | 158 | 157 | 325
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 14 | 11 | 25
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 2 | 1 | 3
    White | 10 | 133 | 141 | 284
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 9 | 4 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 14 | 11 | 25
  Black or African American | 0 | 2 | 1 | 3
  Hispanic or Latino | 0 | 3 | 5 | 8
  Other | 0 | 13 | 9 | 22
  White Non-Hispanic | 10 | 127 | 131 | 268
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 0 | 10 | 18 | 28
  Belgium | 3 | 11 | 6 | 20
  France | 0 | 6 | 2 | 8
  Germany | 0 | 14 | 18 | 32
  Israel | 0 | 18 | 11 | 29
  Italy | 0 | 12 | 11 | 23
  Poland | 0 | 13 | 11 | 24
  Russia | 0 | 30 | 26 | 56
  Spain | 7 | 17 | 19 | 43
  Sweden | 0 | 2 | 0 | 2
  Taiwan, Province Of China | 0 | 8 | 4 | 12
  Turkey | 0 | 2 | 5 | 7
  United Kingdom | 0 | 1 | 3 | 4
  United States | 0 | 10 | 16 | 26
  Korea, Republic Of | 0 | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Part B: Percentage of Participants Who Achieved Complete Response (Complete Response Rate) Based on Investigator Assessment
Description: Complete response rate defined as percentage of participants who achieved complete response as per modified International Working Group (IWG) criteria. CR: Bone marrow blasts less than (<)5 percent (%); absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count greater than (>)1.0*10^9/liter (L) (1000/micro liter [mcL]); platelet count >100*10^9/L (100 000/mcL); independence of red cell transfusions. This endpoint is reported here for Part B only as per the planned analysis.
Time Frame: Approximately up to 2.5 years
Population: Intent-to-Treat (ITT) population is defined as all randomized participants, grouped per treatment assigned by randomization, regardless of the actual treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | Part B: Decitabine (Alone) | Part B: Decitabine + JNJ-56022473
Number analyzed (Participants) | 159 | 157
Percentage of participants | 11.9 | 16.6
Statistical Analysis 1: Comparison: Part B: Decitabine (Alone) vs Part B: Decitabine + JNJ-56022473; Statistical Analysis 1; Test type: Superiority; p = 0.4747, Chi-squared; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.8 to 2.8]

2. Primary Outcome: Part B: Overall Survival
Description: Overall Survival (OS) was defined as the time from the date of randomization to date of death from any cause. Median Overall Survival was estimated by using the Kaplan-Meier method. This endpoint is reported here for Part B only as per the planned analysis.
Time Frame: Approximately up to 2.5 years
Population: ITT population is defined as all randomized participants, grouped per treatment assigned by randomization, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Decitabine (Alone) | Part B: Decitabine + JNJ-56022473
Number analyzed (Participants) | 159 | 157
Months | 7.26 [6.47 to 8.64] | 5.36 [4.27 to 7.95]
Statistical Analysis 1: Comparison: Part B: Decitabine (Alone) vs Part B: Decitabine + JNJ-56022473; Statistical Analysis 1; Test type: Superiority; p = 0.7817, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.79 to 1.37]

3. Secondary Outcome: Part B: Event-free Survival (EFS) Based on Investigator Assessment
Description: EFS defined as time from randomization to treatment failure, relapse from CR/CRi, or death from any cause, whichever occurs first, per modified IWG criteria. Treatment failure: >25% absolute increase in the bone marrow blast count from baseline to present assessment (example, 20% to 46%) on bone marrow aspirate (or biopsy in case of dry tap); Relapse: Bone marrow blasts greater than equal to (>=)5%; reappearance of blasts in blood; or development of extramedullary disease; CR: Bone marrow blasts <5 %; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count > 1.0*10^9/L (1000/mcL); platelet count >100*10^9/L (100 000/mcL);independence of red cell transfusions; CRi: Bone marrow blasts <5 %; absence of blasts with Auer rods; absence of extramedullary disease; residual neutropenia <1.0*10^9/L (1000/mcL) or thrombocytopenia <100*10^9/L (100 000/mcL); independence of red cell transfusions. Endpoint reported is for Part B only as per planned analysis.
Time Frame: Approximately up to 2.5 years
Population: ITT population defined as all randomized participants, grouped per treatment assigned by randomization, regardless of actual treatment received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Decitabine (Alone) | Part B: Decitabine + JNJ-56022473
Number analyzed (Participants) | 159 | 157
Months | 6.24 [4.96 to 6.83] | 4.50 [3.61 to 6.74]

4. Secondary Outcome: Part B: Percentage of Participants Who Achieved CR and CRi (Overall Response Rate)
Description: Percentage of participants who achieved CR and CRi, as per modified IWG criteria. CR: Bone marrow blasts less than (<)5 %; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count greater than (>)1.0 *10^9/liter (L) (1000/ mcL); platelet count >100 *10^9/L (100 000/mcL); independence of red cell transfusions; CRi: Bone marrow blasts <5 %; absence of blasts with Auer rods; absence of extramedullary disease; residual neutropenia <1.0*10^9/L (1000/mcL) or thrombocytopenia <100*10^9/L (100 000/mcL); independence of red cell transfusions. This endpoint is reported here for Part B only as per the planned analysis.
Time Frame: Approximately up to 2.5 years
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Part B: Decitabine (Alone) | Part B: Decitabine + JNJ-56022473
Number analyzed (Participants) | 159 | 157
Percentage of Participants | 20.1 | 26.8

5. Secondary Outcome: Part B: Percentage of Participants With Complete Response (CR) Plus Minimal Residual Disease (MRD) Negative Complete Response With Incomplete Recovery (CRi)
Description: Percentage of participants who achieved CR plus MRD-negative CRi were reported. MRD negativity defined as <1 blast or leukemic stem cell in 10,000 leukocytes (MRD level <10^4).CR: Bone marrow blasts less than (<)5 percent (%); absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count greater than (>)1.0*10^9/liter (L) (1000/mcL); platelet count >100*10^9/L (100 000/mcL); independence of red cell transfusions; CRi: Bone marrow blasts <5 %; absence of blasts with Auer rods; absence of extramedullary disease; residual neutropenia <1.0*10^9/L (1000/mcL) or thrombocytopenia <100*10^9/L (100 000/mcL); independence of red cell transfusions. This endpoint is reported here for Part B only as per the planned analysis.
Time Frame: Approximately 2.5 years
Population: Population included participants in ITT, among whom MRD negativity was evaluated upon achieving response.
Measure: Number; unit: Percentage of participants
Arm/Group | Part B: Decitabine (Alone) | Part B: Decitabine + JNJ-56022473
Number analyzed (Participants) | 80 | 80
Percentage of participants | 13.8 | 21.3

6. Secondary Outcome: Part B: Time to Best Response
Description: Time to best response is calculated as the time from the randomization date to the first documented date for the best response for participants who achieved CR or CRi, as per modified IWG criteria. CR: Bone marrow blasts less than (<)5 %; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count greater than (>)1.0 *10^9/liter (L) (1000/mcL); platelet count >100*10^9/L (100 000/mcL); independence of red cell transfusions; CRi: Bone marrow blasts <5 %; absence of blasts with Auer rods; absence of extramedullary disease; residual neutropenia <1.0*10^9/L (1000/mcL) or thrombocytopenia <100*10^9/L (100 000/mcL); independence of red cell transfusions. This endpoint is reported here for Part B only as per the planned analysis.
Time Frame: Approximately 2.5 years
Population: Population included participants in ITT, who achieved CR or CRi.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Part B: Decitabine (Alone) | Part B: Decitabine + JNJ-56022473
Number analyzed (Participants) | 32 | 42
Weeks | 16.71 [7.1 to 41.6] | 18.14 [7.3 to 68.4]

7. Secondary Outcome: Part B: Duration of Response (DOR) Based on Investigator Assessment
Description: DOR defined as number of weeks from documented best response (CR or CRi) for participants who achieved CR or CRi to relapse, death due to relapse, date of censoring. As per modified IWG criteria: CR: Bone marrow blasts <5 %; absence of blasts with Auer rods; absence of extramedullary disease;absolute neutrophil count >1.0*10^9/L (1000/mcL); platelet count >100*10^9/L (100 000/mcL); independence of red cell transfusions; CRi: Bone marrow blasts <5 %; absence of blasts with Auer rods; absence of extramedullary disease; residual neutropenia <1.0* 10^9/L (1000/mcL) or thrombocytopenia <100*10^9/L (100 000/mcL); independence of red cell transfusions. This endpoint is reported here for Part B only as per the planned analysis.
Time Frame: Approximately 2.5 years
Population: Population included participants in ITT, who achieved CR or CRi.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Part B: Decitabine (Alone) | Part B: Decitabine + JNJ-56022473
Number analyzed (Participants) | 32 | 42
Weeks | 23.71 [15.43 to NA] — Upper limit of 95% confidence interval (CI) was not estimable due to insufficient number of events. | NA [29.86 to NA] — Median and upper limit of 95% CI was not estimable due to insufficient number of events.

ADVERSE EVENTS:
Time Frame: Throughout the study (Up to 2.5 years)
Description: Safety Population defined as randomized participants who received at least one dose of study medication, grouped according to actual treatment received (9 participants from decitabine + JNJ-56022473 arm were grouped in the decitabine alone arm as they received only decitabine and not JNJ 56022473). All-cause mortality is reported here for randomized participants. Serious and Other (Not including Serious) Adverse Events are reported for Safety Population per planned analysis.
Arm/Group | Part A: Decitabine + JNJ-56022473 | Part B: Decitabine (Alone) | Part B: Decitabine + JNJ-56022473
All-Cause Mortality (participants affected / at risk) | 10/10 | 101/159 | 99/157
Serious Adverse Events (participants affected / at risk) | 9/10 | 120/165 | 126/147
Other Adverse Events (participants affected / at risk) | 9/10 | 157/165 | 146/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Decitabine + JNJ-56022473 (N=10) | Part B: Decitabine (Alone) (N=165) | Part B: Decitabine + JNJ-56022473 (N=147)
Anaemia (Blood and lymphatic system disorders) | 0 | 6 | 4
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 1 | 1
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 36 | 40
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2 | 2
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 5 | 3
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 3
Angina Pectoris (Cardiac disorders) | 0 | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 2 | 5
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1 | 5
Cardiac Failure (Cardiac disorders) | 0 | 2 | 0
Cardiac Failure Acute (Cardiac disorders) | 0 | 2 | 0
Cardiogenic Shock (Cardiac disorders) | 0 | 1 | 0
Cardiopulmonary Failure (Cardiac disorders) | 0 | 1 | 1
Cardiovascular Insufficiency (Cardiac disorders) | 0 | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 1 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 3
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0
Acute Abdomen (Gastrointestinal disorders) | 0 | 1 | 0
Anal Ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 2
Diverticular Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum Intestinal (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis Erosive (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Angiodysplasia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Polyp Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Mechanical Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 3
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 2
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Asthenia (General disorders) | 0 | 0 | 3
Catheter Site Inflammation (General disorders) | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 3
Death (General disorders) | 0 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 3
General Physical Health Deterioration (General disorders) | 1 | 6 | 4
Hyperthermia (General disorders) | 0 | 0 | 1
Influenza Like Illness (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 2
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 9 | 9
Pyrexia (General disorders) | 1 | 9 | 15
Sudden Death (General disorders) | 0 | 5 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis Acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic Reaction (Immune system disorders) | 0 | 1 | 1
Anaphylactic Shock (Immune system disorders) | 0 | 0 | 2
Serum Sickness (Immune system disorders) | 0 | 0 | 1
Actinomycotic Pulmonary Infection (Infections and infestations) | 0 | 1 | 0
Alveolar Osteitis (Infections and infestations) | 0 | 0 | 1
Anal Infection (Infections and infestations) | 0 | 1 | 0
Aspergillus Infection (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 2 | 1
Bacterial Sepsis (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 2
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 | 1 | 0
Candida Infection (Infections and infestations) | 0 | 1 | 0
Catheter Site Infection (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 2 | 3
Clostridial Infection (Infections and infestations) | 0 | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 1
Clostridium Difficile Infection (Infections and infestations) | 0 | 1 | 0
Device Related Infection (Infections and infestations) | 2 | 3 | 3
Device Related Sepsis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Enterobacter Bacteraemia (Infections and infestations) | 0 | 0 | 1
Escherichia Bacteraemia (Infections and infestations) | 0 | 0 | 3
Escherichia Infection (Infections and infestations) | 0 | 0 | 1
Escherichia Sepsis (Infections and infestations) | 2 | 0 | 2
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Fungaemia (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis Rotavirus (Infections and infestations) | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1
Gastrointestinal Candidiasis (Infections and infestations) | 0 | 1 | 0
Hepatic Infection Fungal (Infections and infestations) | 0 | 1 | 1
Infected Skin Ulcer (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 3
Infectious Colitis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 1
Klebsiella Infection (Infections and infestations) | 0 | 0 | 2
Liver Abscess (Infections and infestations) | 0 | 2 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 1
Lung Infection (Infections and infestations) | 4 | 5 | 3
Meningitis (Infections and infestations) | 0 | 0 | 1
Moraxella Infection (Infections and infestations) | 0 | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 0 | 1 | 1
Oral Candidiasis (Infections and infestations) | 0 | 1 | 0
Parainfluenzae Virus Infection (Infections and infestations) | 0 | 1 | 1
Parotitis (Infections and infestations) | 0 | 1 | 0
Periorbital Cellulitis (Infections and infestations) | 0 | 1 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 23 | 24
Pneumonia Fungal (Infections and infestations) | 0 | 1 | 1
Pseudomembranous Colitis (Infections and infestations) | 0 | 0 | 1
Pulmonary Mycosis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 1
Pyelonephritis Chronic (Infections and infestations) | 0 | 0 | 1
Rash Pustular (Infections and infestations) | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 4
Rhinovirus Infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 2 | 6 | 14
Septic Encephalopathy (Infections and infestations) | 0 | 1 | 0
Septic Shock (Infections and infestations) | 0 | 2 | 8
Sinusitis Fungal (Infections and infestations) | 0 | 0 | 1
Skin Infection (Infections and infestations) | 1 | 1 | 1
Splenic Abscess (Infections and infestations) | 0 | 1 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 0 | 0 | 2
Tooth Abscess (Infections and infestations) | 0 | 0 | 1
Tooth Infection (Infections and infestations) | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 4 | 6
Urosepsis (Infections and infestations) | 0 | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1 | 0
Vulval Cellulitis (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 4
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Transfusion Reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Transfusion-Related Acute Lung Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 1
C-Reactive Protein Increased (Investigations) | 0 | 1 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Central Nervous System Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 3
Dizziness (Nervous system disorders) | 0 | 2 | 2
Epilepsy (Nervous system disorders) | 0 | 1 | 1
Haemorrhage Intracranial (Nervous system disorders) | 0 | 1 | 0
Haemorrhagic Stroke (Nervous system disorders) | 0 | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Quadriparesis (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 4
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1 | 1
Vascular Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 4
Anuria (Renal and urinary disorders) | 0 | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Respiratory Tract Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash Vesicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 3
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 2
Phlebitis (Vascular disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Condition Aggravated (General disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemodynamic Instability (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Decitabine + JNJ-56022473 (N=10) | Part B: Decitabine (Alone) (N=165) | Part B: Decitabine + JNJ-56022473 (N=147)
Anaemia (Blood and lymphatic system disorders) | 7 | 80 | 77
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 22 | 25
Leukocytosis (Blood and lymphatic system disorders) | 0 | 9 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 15 | 12
Neutropenia (Blood and lymphatic system disorders) | 1 | 61 | 64
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 86 | 81
Atrial Fibrillation (Cardiac disorders) | 0 | 8 | 13
Tachycardia (Cardiac disorders) | 1 | 6 | 14
Abdominal Pain (Gastrointestinal disorders) | 1 | 12 | 19
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 6 | 9
Anal Incontinence (Gastrointestinal disorders) | 0 | 0 | 10
Constipation (Gastrointestinal disorders) | 3 | 51 | 47
Diarrhoea (Gastrointestinal disorders) | 4 | 41 | 50
Dyspepsia (Gastrointestinal disorders) | 1 | 5 | 10
Gingival Bleeding (Gastrointestinal disorders) | 0 | 10 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 8 | 21
Nausea (Gastrointestinal disorders) | 5 | 33 | 36
Stomatitis (Gastrointestinal disorders) | 1 | 16 | 12
Toothache (Gastrointestinal disorders) | 0 | 9 | 4
Vomiting (Gastrointestinal disorders) | 5 | 19 | 26
Asthenia (General disorders) | 2 | 25 | 26
Chills (General disorders) | 3 | 7 | 30
Fatigue (General disorders) | 1 | 31 | 31
Oedema Peripheral (General disorders) | 5 | 25 | 46
Pain (General disorders) | 0 | 5 | 8
Pyrexia (General disorders) | 6 | 46 | 51
Oral Candidiasis (Infections and infestations) | 2 | 6 | 9
Oral Herpes (Infections and infestations) | 3 | 9 | 11
Pneumonia (Infections and infestations) | 1 | 19 | 19
Urinary Tract Infection (Infections and infestations) | 0 | 13 | 13
Contusion (Injury, poisoning and procedural complications) | 0 | 5 | 8
Fall (Injury, poisoning and procedural complications) | 0 | 9 | 13
Alanine Aminotransferase Increased (Investigations) | 0 | 5 | 9
Aspartate Aminotransferase Increased (Investigations) | 0 | 5 | 8
Blood Creatinine Increased (Investigations) | 0 | 4 | 8
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 1 | 8
Weight Decreased (Investigations) | 0 | 10 | 16
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 31 | 25
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 17
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 8 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 5 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 9 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 41 | 53
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 12 | 20
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 5 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 15 | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 18 | 19
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 12 | 15
Dizziness (Nervous system disorders) | 1 | 9 | 14
Headache (Nervous system disorders) | 1 | 15 | 16
Insomnia (Psychiatric disorders) | 2 | 13 | 16
Acute Kidney Injury (Renal and urinary disorders) | 0 | 7 | 11
Urinary Incontinence (Renal and urinary disorders) | 0 | 5 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 15 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 23 | 22
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 13 | 20
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 8
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 9
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 10 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 4 | 9
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 10 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 12 | 11
Rash (Skin and subcutaneous tissue disorders) | 1 | 11 | 13
Hypertension (Vascular disorders) | 0 | 13 | 24
Hypotension (Vascular disorders) | 1 | 17 | 22
Syncope (Nervous system disorders) | 2 | 5 | 6
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 7
Splenomegaly (Blood and lymphatic system disorders) | 1 | 2 | 2
Tympanic Membrane Disorder (Ear and labyrinth disorders) | 1 | 0 | 0
Uveitis (Eye disorders) | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 1 | 6
Parotid Gland Enlargement (Gastrointestinal disorders) | 1 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gait Disturbance (General disorders) | 2 | 0 | 1
General Physical Health Deterioration (General disorders) | 1 | 2 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 7 | 3
Bronchitis (Infections and infestations) | 1 | 5 | 5
Lung Infection (Infections and infestations) | 1 | 4 | 2
Lymph Gland Infection (Infections and infestations) | 1 | 0 | 0
Oropharyngeal Candidiasis (Infections and infestations) | 1 | 0 | 2
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 3
Skin Infection (Infections and infestations) | 1 | 3 | 2
Systemic Mycosis (Infections and infestations) | 1 | 0 | 0
Tooth Abscess (Infections and infestations) | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 6 | 2
Bacterial Test Positive (Investigations) | 1 | 0 | 1
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 0
International Normalised Ratio Increased (Investigations) | 1 | 3 | 4
Oxygen Saturation Decreased (Investigations) | 1 | 0 | 4
Fluid Overload (Metabolism and nutrition disorders) | 1 | 4 | 6
Fluid Retention (Metabolism and nutrition disorders) | 1 | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 4 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 7 | 4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4
Somnolence (Nervous system disorders) | 1 | 2 | 2
Adjustment Disorder with Depressed Mood (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 3 | 4
Depressed Mood (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 2 | 1
Nervousness (Psychiatric disorders) | 1 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 3 | 5
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 3 | 2
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/45/NCT02472145/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT02472145/SAP_001.pdf